CLINICAL TRIAL: NCT03817905
Title: Incomplete Follow Up After Positive FIT or Stool DNA Testing: A Multimethod Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1219
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Positive FIT or Stool DNA Testing Follow up
Keywords: Colonoscopy; Fecal Immunochemical Testing
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient navigator (Experimental): Participant meets the patient navigator at their colonoscopy appointment and discusses any problems they experienced in getting the colonoscopy done. Participant will tell navigator in their own words their experience and whether they faced any barriers to scheduling and colonoscopy completion.
  Interventions: Other: Patient navigator

INTERVENTIONS:
Other: Patient navigator — Intervention will utilize staff at the Seidman Cancer Center who are trained in patient navigation and have experience in navigating patients for breast cancer screening as well as sickle cell disease. The staff will undergo training for this study by study principal investigators which will include the target participant population, necessary steps in the navigation process and data that will be collected. In addition, they will receive brief training in supportive, listening technique. They will also be furnished with a telephone script for the initial participant contact.

SUMMARY:
This study seeks to determine whether a patient navigator can help improve follow up care after a stool test shows the presence of blood or other abnormal markers.

DETAILED DESCRIPTION:
Participants who recently had a stool test that had abnormal results will be asked to participate in this study in order to determine whether the use of a navigator can increase the use of colonoscopy, which is the recommended follow up to an abnormal stool test. A navigator is an individual trained to help patients access necessary health care services and understand the test results and next steps. Participants will be asked to meet the navigator at their colonoscopy appointment and discuss any problems that are experienced in getting the colonoscopy done. This will take about 10 minutes to complete. Participants will tell him or her in their own words how the experience was and whether they faced any barriers to scheduling and colonoscopy completion. Study personnel will also look at participants' electronic medical record to see what testing participants had done that prompted the need for colonoscopy.The study will include about 30 people.

ELIGIBILITY:
Inclusion Criteria:

• Positive test for FIT or sDNA

Exclusion Criteria:

• Does not understand English

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants completing a follow-up colonoscopy procedure | Up to 6 months from start of study
  Feasibility of a navigator based intervention to improve follow up will be determined by comparing the colonoscopy completion rate to historical controls. This will be measured as number of participants completing a follow-up colonoscopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cooper, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States